CLINICAL TRIAL: NCT01373944
Title: Rapid-Acquisition Low-Dosimetry Tc-99m Stress-Only Myocardial Perfusion SPECT on the Spectrum Dynamics System: Comparison of Efficiency and Outcomes With Stress-Only Anger SPECT
Brief Title: Efficiency and Outcomes of Stress-Only Anger and D-SPECT Stress-Only SPECT MPI
Status: Completed | Type: Observational
Sponsor: Aspire Foundation (Other)
Collaborators: Spectrum Dynamics (Industry); Cardiovascular Imaging Technologies, LLC (Unknown); Saint Luke's Cardiovascular Consultants (Other); Mid America Heart Institute (Other)
Responsible Party: Timothy M. Bateman, MD, Medical Director, Aspire Foundation
Other Study IDs: D-Spect Stress Only
Record Dates: First submitted 2011-06-14; First posted 2011-06-15 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Coronary Artery Disease
Keywords: MPI; SPECT; Stress-Only; Spectrum Dynamics Camera; Anger
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stress Only SPECT MPI with Anger Camera: Patients undergoing clinically-indicated stress-only sestamibi studies who are imaged on the traditional Anger camera
- Stress Only SPECT MPI with SD Camera: Patients undergoing clinically-indicated stress-only sestamibi studies who are imaged on the Spectrum Dynamics camera system.

SUMMARY:
The purpose of this study is to compare clinical efficiency and patient outcomes using ultra low-dose stress only Tc-99m and solid-state SPECT versus traditional Anger SPECT.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 35 kg/m2
* LVEF > 40%
* Exercise stress
* Elective out-patients
* No known CAD (>50%) by catheterization
* No history of prior myocardial infarction

Exclusion Criteria:

* LBBB
* Pacemaker
* Atrial Fibrillation
* Frequent PAC's or PVC's
* Inability to achieve at least 6 minutes

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred for clinically-indicated myocardial perfusion SPECT
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic Failure | 30 days
  Diagnostic failure is defined by a composite of need for additional downstream testing (anger SPECT, MPI PET, stress echocardiography or coronary CT angiography) within 30 days or a coronary angiogram with no stenoses greater than or equal to 50% severity using quantitative coronary angiography.

SECONDARY OUTCOMES:
Necessity to proceed to a rest image | 30 days
  The first of 4 secondary end-points is the need to proceed to a rest image.
Necessity for additional downstream testing | 30 days
  The second of four secondary endpoints the need for additional downstream testing within 30 days to address the same clincial reason for the innitial referral for stress-onoly imaging, in the absence of any changes in clincial status between tests.
Coronary Angiography | 60 to 90 days
  The third of four secondary end-points is the occurrence of coronary angiography with no stenoses greater than or equal to 50% severity using quantitative coronary angiography.
Determine optimal performance of the Spectrum Dynamics camera system for stress only imaging | 60 to 90 days
  The fourth of four secondary endpoints is to determine optimal performance of the Spectrum Dynamics camera system for stress only imaging: upright imaging alone, supine imaging alone, or both in terms of primary and secondary endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Bateman, MD, Principal Investigator — Aspire Foundation
Locations (3):
- United States (3):
  - Saint Luke's Cardiovascular Imaging Center, Kansas City, Missouri
  - Saint Luke's North Cardiovascular Imaging Center, Kansas City, Missouri
  - Saint Luke's East Cardiovascular Imaging Center, Lee's Summit, Missouri